CLINICAL TRIAL: NCT04643535
Title: Glycocalyx as Predictor of Complications After Cardiac Surgery
Brief Title: In Vivo Glycocalyx as Predictor of Complications After Cardiac Surgery
Acronym: GLYPOCS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/202/OB
Record Dates: First submitted 2020-11-19; First posted 2020-11-25 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-11

CONDITIONS: Endothelial Dysfunction; Cardiovascular Diseases; Surgery
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiac surgery has been described as altering endothelium structure and function, notably because of the use of cardiac-pulmonary bypass (CPB). Among the endothelial structure, glycocalyx, the thin layer recovering the endothelial surface, may be altered by the inflammatory process and probably the modification of flow during CPB. Endothelial and glycocalyx integrity are essential for vascular function and glycocalyx destruction is associated with organ failure and mortality. On the other hand, a chronic alteration of glycocalyx is observed in many diseases such as diabetes, hypertension or chronic kidney failure, all pathologies frequently observed in patients benefiting grom cardiac surgery.

Thus the preoperative alteration of glycocalyx may be associated with postoperative organ failure.

ELIGIBILITY:
Inclusion Criteria:

* all patients benefiting from a cardiac surgery with cardio-pulmonary bypass

Exclusion Criteria:

* impossibility to carry out the measurement by glycocheck device
* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients benefiting from cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
association between preoperative sublingual glycocalyx thickness (glycocheck device) and major postoperative complications | 48 hours
  occurence within 48 postoperative hours of at least one item among:
  * vasoplegic shock
  * cardiogenic shock
  * prolonged mechanical ventilation
  * acute kidney failure
  * Death

SECONDARY OUTCOMES:
association between preoperative sublingual glycocalyx thickness (glycocheck device) and death | 28 days
  death from any causes
association between preoperative sublingual glycocalyx thickness (glycocheck device) and cardiac arrythmia | 28 days
  atrial or ventricular arrythmia
association between preoperative sublingual glycocalyx thickness (glycocheck device) and Cerebral stroke | 28 days
  ischemic of hemorrhagic etiology
association between preoperative sublingual glycocalyx thickness (glycocheck device) and cognitive dysfunction | 28 days
  delirium or alteration of cognitive status
association between preoperative sublingual glycocalyx thickness (glycocheck device) and myocardial ischemia | 28 days
  occurence of ischemia: new Q wave, new occlusion of a coronary arteria, elevated troponinemia with a new dysfunction of at least one myocardial segment
association between preoperative sublingual glycocalyx thickness (glycocheck device) and acute respiratory failure | 28 days
  need for at least 5L/min of oxygen or non invasive ventilation of reintubation
association between preoperative sublingual glycocalyx thickness (glycocheck device) and sepsis | 28 days
  new sepsis condition as defined by SEPSIS-3 definition

CONTACTS AND LOCATIONS:
Locations (1):
- Rouen University Hospital, Rouen, France